CLINICAL TRIAL: NCT02237105
Title: The Effect of Cognitive Behavioral Therapy on the Outcome of Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC14276-13CTIL
Record Dates: First submitted 2014-06-08; First posted 2014-09-11 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy Group (Experimental): This group will undergo Cognitive Behavioral Therapy (CBT) before having spinal surgery
  Interventions: Behavioral: Cognitive Behavioral Therapy
- control group (No Intervention): This group will not undergo any psychological intervention before the spinal surgery.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy
  Arms: Cognitive Behavioral Therapy Group

SUMMARY:
This study is designed to examine the efficacy of Cognitive Behavioral Therapy (CBT) on the outcome of spinal surgery.

The goal of this treatment is to change the coping style, thoughts, behavior and adaptive perception of the patient, and to replace them with an adaptive style.

The patients in this study will be randomly divided into two groups. One group will undergo Cognitive Behavioral Therapy (CBT) before having spinal surgery. The other group will be a control group, and will not have any psychological intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients who intended to undergo spinal surgery

Exclusion Criteria:

* patients who does not speak Hebrew language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
BSI questionnaire in spine preoperative patients . | 24 months
  assessment of emotional state in spine preoperative patients will be measured by analysis of BSI questionnaire
OSWESTRY questionnaire in spine preoperative patients | 24 months
  Assessment of disability in spine preoperative patients will be measured by analysis of OSWESTRY questionnaire
SF 36 questionnaire in spine preoperative patients | 24 months
  assessment of well being in preoperative patients will be measured by analysis of SF36 questionnaire
VAS scale in spine preoperative patients | 24 months
  Assessment of pain intensity in spine preoperative patients will be measured by analysis of VAS scale

SECONDARY OUTCOMES:
BSI questionnaire in spine postoperative patients | 24 months
  assessment of emotional state in spine postoperative patients will be measured by analysis of BSI questionnaire
OSWESTRY questionnaire in spine postoperative patients | 24 months
  Assessment of disability in spine postoperative patients will be measured by analysis of OSWESTRY questionnaire
SF 36 questionnaire in postoperative patients | 24 months
  Assessment of well being in spine postoperative patients will be measured by analysis of SF 36 questionnaire
VAS scale in spine postoperative patients | 24 months
  Assessment of pain intensity in spine postoperative patients will be measured by analysis of VAS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Meir MC, Kfar Saba, Israel